CLINICAL TRIAL: NCT04535115
Title: Intraoperative Hemodynamic Optimization: Predictive Value to Fluid Respon-siveness of the Tidal Volume Challenge and the Lung Recruitment Maneuver by Monitoring the Variation of the Pulsed Pressure and the Variation of the Systolic Ejection Volume.
Brief Title: Tidal Volume Challenge and Lung Recruitment Maneuver (TIDALREC): the Reliability of Pulse Pression Variation or Stroke Volume Variation on Fluid Responsiveness.
Acronym: TIDALEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019_71; 2020-A01460-39 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Fluid Challenge; Hemodynamic Monitoring
Keywords: Tidal Volume Challenge; Lung Recruitment Maneuver; Pulse Pression Varia-tion; Stroke Volume Variation.; Fluid Responsiveness.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Starting LRM (Lung Recruitment Maneuver)
  Interventions: Procedure: Starting LRM (Lung Recruitment Maneuver)
- Group 2 (Experimental): Starting VtC (Tidal Volume Challenge)
  Interventions: Procedure: Starting VtC (Tidal Volume Challenge)

INTERVENTIONS:
Procedure: Starting LRM (Lung Recruitment Maneuver) — The LRM is performed first for 30 seconds (an insufflation pressure of 30 cmH2O for 30 seconds is applied). After a free interval of 3 minutes, the VtC is done during 1 minute. For VtC, tidal volume is increased from 6 to 8 ml.kg-1 of predicted body weight. Finally, after a new free interval of 3 minutes, the fluid challenge (consisting in fluid administration of 250 ml of Ringer Lactate) is started for 10 minutes (in aim to determine which patients are responders). This sequence is repeated every 30 minutes (maximum four times).
  Arms: Group 1
Procedure: Starting VtC (Tidal Volume Challenge) — The VtC is performed first for 1 minute. After a free interval of 3 minutes, the LRM is done for 30 seconds. Finally, after another free interval of 3 minutes, the fluid challenge is started for 10 minutes. This sequence is repe-tead every 30 minutes (maximum four times).
  Arms: Group 2

SUMMARY:
In order to predict fluid responsiveness in the operating room and therefore benefit of performing fluid administration to improve patient's hemodynamic status, it will test two ventilation strategies : the Tidal Volume Challenge (VtC) and the Lung Recruitment Maneuver (LRM).

The objective is to determine whether the variation of 2 parameters such as pulse pression variation (PPV) and stroke volume variation (SVV) during these 2 strategies, allows to predict fluid responsiveness in the operating room for any heavy surgery. All patients will benefit from the 2 ventilation strategies then a fluid administration, called " fluid challenge ", will be performed to discriminate the true responders and others. The order of the ventilation strategies will be determined by randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major abdominal, vascular or neurosurgery requiring invasive arterial monitoring of SVV and PPV with placement of a radial arterial catheter connected to the ProAQT® System.
* Block duration > 2 hours.

Exclusion Criteria:

* open surgery
* history of supra ventricular arrhythmias
* beta-blocking patient
* BMI>30 kg.m-2 or <15 kg.min-2
* right ventricular dysfunction
* severe valvulopathies
* intracardiac shunt
* renal failure dialysis
* patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
The area under the ROC curve (AUC) of the variation of the pulsed pressure (VPP) during the tidal volume challenge (VtC). | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 30 minutes that can occur several times during surgery

SECONDARY OUTCOMES:
The area under the ROC (AUC) curve of VPP during the alveolar recruit-ment maneuver. | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 30 minutes that can occur several times during surgery
  The AUCs are measured before and after each strategies. Afterwards, the measurement is done before and after the " fluid challenge " in each group. This sequence of measurements will be recorded every 30 minute
The AUCs of the two techniques calculated above. | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 30 minutes that can occur several times during surgery
  The AUCs are measured before and after each strategies. Afterwards, the measurement is done before and after the " fluid challenge " in each group. This sequence of measurements will be recorded every 30 minute
The area under the ROC curve (AUC) of stroke volume variation (SVV) during the tidal volume challenge (VtC). | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 30 minutes that can occur several times during surgery
  The AUCs are measured before and after each strategies. Afterwards, the measurement is done before and after the " fluid challenge " in each group. This sequence of measurements will be recorded every 30 minute
The area under the ROC curve (AUC) of stroke volume variation (SVV) during the lung recruitment maneuver. | throughout surgery (mean length expected between 3 and 5 hours). Measurements performed during sequences of 30 minutes that can occur several times during surgery
  The AUCs are measured before and after each strategies. Afterwards, the measurement is done before and after the " fluid challenge " in each group. This sequence of measurements will be recorded every 30 minute
Number of complications in pneumothorax | 1 day (at recovery room after surgery) and at day 2
  Pneumothorax is detected on chest x-ray in recovery room and then on clinical examination at Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France